CLINICAL TRIAL: NCT05188924
Title: A Multi-center, Randomized, Double-blinded, Placebo-controlled Clinical Trial to Evaluate the Efficacy and Safety of DKF-306 in Patients With Periodontal Diseases
Brief Title: Efficacy and Safety of DKF-306 in Patients With Periodontal Diseases
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dongkook Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DKF-306-P4
Record Dates: First submitted 2021-12-27; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DKF-306 (Experimental): During Weeks 1 to 4, 2 tablets, t.i.d. During Weeks 5 to 12, 1 tablet, t.i.d.
  Interventions: Drug: DKF-306
- Placebo (Placebo Comparator): During Weeks 1 to 4, 2 tablets, t.i.d. During Weeks 5 to 12, 1 tablet, t.i.d.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DKF-306 — Active ingredients
  Arms: DKF-306
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double-blinded, placebo-controlled study to evaluated the efficacy and safety of DKF-306 in patients with periodontal diseases.

ELIGIBILITY:
Inclusion Criteria:

* Aged 19 years and older
* Periodontal diseases
* Having not less than 16 permanent teeth including at least 4 molars (third molars excluded)
* Having teeth with not less than 2 sites of both probing pocket depth (PPD) ≥ 4 mm and gingival index (GI) ≥ 2 in at least 2 quadrants
* Agrees not to use over-the-counters (oral, ointment, toothpaste, film, etc.) or quasi-drugs (gargle and mouthwash) to alleviate or treat the symptoms of gingivitis or periodontitis during the study
* Voluntarily signed the informed consent form
* Willing to participate in the study

Exclusion Criteria:

* Hypersensitivity to ingredients of investigational products
* Hypersensitivity to Azo dyes, acetylsalicylic acid or other prostaglandin synthase inhibitors
* Following diseases or state in the mouth:

  1. rampant caries or decayed tooth/teeth remained untreated for a long time
  2. multiple restorations which may be related to periodontal inflammation
  3. poor oral hygiene with heavy plaque or calculus deposition
  4. soft or hard tissue tumor
  5. systemic chronic diseases with oral manifestations
  6. fibrotic gingival enlargement
* Use of orthodontic appliances or removable partial denture(s)
* Having teeth or state in need of immediate treatment such as periodontal abscess, a tooth indicated for extraction, etc.
* History of aggressive periodontitis or acute necrotizing ulcerative gingivitis
* Received dental treatments such as endodontic treatments or periodontal therapy (including both nonsurgical and surgical therapy) within 3 months from randomization
* Received the following drugs for more than 2 weeks within 3 months from randomization:

  1. systemic/local antibiotics in the mouth or non-steroidal anti-inflammatory drugs
  2. cyclosporine or corticosteroids
  3. phenytoin, calcium antagonists, anticoagulants or antiplatelets
* Initiated drugs in treatment of chronic diseases within 3 months from randomization
* Received the same drug with investigational products within 3 months from randomization
* Medical conditions or diseases affecting the efficacy and safety of investigational products at the investigator's discretion
* Heavy smoker (20 cigarettes or more a day)
* Pregnant or breast-feeding
* Plans to have a child or unwilling to comply with using medically accepted contraception methods during the study
* Alcohol or drug abuse
* Other investigational products or procedures within 3 months from screening
* Not eligible due to other reasons at the investigator's discretion

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2020-05-22 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in gingival index from baseline to Week 12 | Weeks 0 and 12

SECONDARY OUTCOMES:
Change in plaque index from baseline to Weeks 4, 8 and 12 | Weeks 0, 4, 8 and 12
Change in probing pocket depth from baseline to Weeks 4, 8 and 12 | Weeks 0, 4, 8 and 12
Change in clinical attachment level from baseline to Weeks 4, 8 and 12 | Weeks 0, 4, 8 and 12
Change in bleeding on probing (%) from baseline to Weeks 4, 8 and 12 | Weeks 0, 4, 8 and 12
Change in gingival index from baseline to Weeks 4 and 8 | Weeks 0, 4 and 8

CONTACTS AND LOCATIONS:
Locations (1):
- Youngsung, Seoul, South Korea